CLINICAL TRIAL: NCT05558150
Title: A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interactions and Safety After Co-administration of Ilaprazole and Aceclofenac in Healthy Adults
Brief Title: Study to Evaluate Pharmacokinetic Drug Interactions and Safety of Ilaprazole and Aceclofenac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REIL49NS01
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — ilaprazole; aceclofenac

STUDY DESIGN:
Intervention Model Description: Randomization, Open-label, Repeated administration, Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ilaprazole & aceclofenac 1 (Experimental): Period 1 : Ilaprazole 10mg/tab, one a day, 5 days
  Period 2 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Period 3 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac
- ilaprazole & aceclofenac 2 (Experimental): Period 1 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Period 2 : Ilaprazole 10mg/tab, one a day, 5 days
  Period 3 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac
- ilaprazole & aceclofenac 3 (Experimental): Period 1 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Period 2 : Period 3 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Period 3 : Ilaprazole 10mg/tab, one a day, 5 days
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac
- ilaprazole & aceclofenac 4 (Experimental): Period 1 : Ilaprazole 10mg/tab, one a day, 5 days
  Period 2 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Period 3 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac
- ilaprazole & aceclofenac 5 (Experimental): Period 1 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Period 2 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Period 3 : Ilaprazole 10mg/tab, one a day, 5 days
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac
- ilaprazole & aceclofenac 6 (Experimental): Period 1 : aceclofenac 100mg/tab, twice a day, 4 days and aceclofenac 100mg/tab, one a day one at the 5 day
  Period 2 : Ilaprazole 10mg/tab, one a day, 5 days
  Period 3 : Ilaprazole 10mg/tab, one a day, 5 days + aceclofenac 100mg/tab, twice a day, 5 days
  Interventions: Drug: Ilaprazole; Drug: Aceclofenac

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 10mg
  Other Names: Noltec(the brand name)
Drug: Aceclofenac — Aceclofenac 100mg
  Other Names: Airtal(the brand name)

SUMMARY:
This study evaluate the pharmacokinetic drug interactions and safety after co-administration of ilaprazole and Aceclofenac in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 or older and 55 or younger at the time of screening tests.
2. Men weigh more than 55 kg and women weigh more than 50 kg.
3. Those who have a body mass index of 18.5 kg/m2 or more and less than 27.0 kg/m2.

   ※ Body mass index (kg/m2) = Weight (kg)/[Height (m)]2
4. If participants are a woman, participants must apply to one of the following.

   * Menopausal (no natural menstruation for at least 2 years)
   * Surgical infertility (autonomous exudation or bilateral ovarian resection, intubation ligation, or other infertility)
5. Men who have sexual relationship with women of child bearing potential must give consent to using contraceptive measures(condoms, spermicide, and menstrual cycle control) for at least 28 days after the final administration of clinical trial and clinical drugs (if the male test subject or female partner is infertile, the above contraception is unnecessary).
6. A person who has heard sufficient explanation of this clinical trial and fully understood it, voluntarily decided to participate, and agreed in writing to comply with precautions.

Exclusion Criteria:

1. A person with a history of mental illness or illness corresponding to clinically significant hepatobiliary tract (hepatic liver disorder, kidney (severe renal disorder, etc.), nervous system, immune system, respiratory system (bronchial asthma, etc.), urinary system, digestive system, endocrine blood and tumor, cardiovascular system (severe high blood pressure, heart failure, etc.).
2. Active peptic ulcer/bleeding or a person with a medical history.
3. A person who tends to bleed or have a blood clotting disorder.
4. Patients with a history of gastrointestinal bleeding or perforation due to NSAID treatment in the past.
5. Those with a history of gastrointestinal diseases (Crohn's disease, ulcerative colitis, etc.) or surgery (except for simple appendectomy or hernia surgery) that can affect the absorption of drugs.
6. Person with a history of significant drug hypersensitivity reactions to the ingredients and additives of clinical trial drugs. In particular, NSAIDs and aspirin such as Yellow No. 4 (Tartrazine), Yellow No. 5 (Sunset Yellow FCF), sulfonamide, ilaprazole and naproxen, aceclofenac, celecoxib, diclofenac, etc.
7. A person with a history of asthma, rhinitis, and nasal polyps due to aspirin or other NSAIDs (including COX-2 inhibitors).
8. A person who was judged to be inappropriate as a test subject in a screening test conducted within 28 days before the first administration date of the clinical trial drug.

   * In the case of > 1.25 times the upper limit of AST and ALT normal range in the blood,
   * When the potassium concentration in the blood exceeds 5.5 mEq/L,
   * Estimated Global Film Rate (eGFR) <60 mL/min/1.73 m2 using the Modification of Diet in Regular Disease (MDRD) formula
   * Immunology and serology tests (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test) result are positive factors.
   * After resting for more than 5 minutes, systolic blood pressure >150 mmHg or << in vital signs measured at the seat> Those who showed values corresponding to 90 mmHg, dilator blood pressure >100 mmHg, or <50 mmHg.
9. A person who has a history of drug abuse or has tested positive in a urine drug screening test within one year of screening.
10. If the tester determines that the following drugs, excluding topical drugs without significant systemic absorption, may affect this test or affect the safety of the test subject within the relevant period,

    * In the case of taking a prescription drug or herbal medicine within 14 days prior to the first administration date of the clinical trial drug,
    * In the case of taking general medicines including health foods and vitamin preparations within 7 days prior to the first administration of clinical trial drugs,
    * A person who took drugs such as barbital drugs and other drugs inducing and inhibiting drugs within 30 days prior to the first administration of clinical trial drugs.
11. A person who continuously smoked excessively or consumed caffeine or alcohol (caffeine: >5 cups/day, alcohol: >210 g/week, tobacco: >10 g/day) or who cannot stop smoking, caffeine and alcohol consumption during each hospitalization period.
12. A person who has consumed grapefruit-containing food within 7 days prior to the first administration date of clinical trial drugs or cannot be prohibited from taking it during the clinical trial period.
13. A person who participated in another clinical trial within 180 days prior to the first administration date of the clinical trial drug and received the clinical trial drug (in the case of biological agents, it may be based on an extended period considering a half-life).
14. A person who donated whole blood within 60 days prior to the first administration date of clinical trial drugs or donated component blood within 30 days.
15. A person who received a blood transfusion within 30 days prior to the first administration date of the clinical trial drug.
16. Pregnant or lactating women.
17. A person who determines that the tester is inappropriate to participate in clinical trials due to other reasons.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
ilaprazole, aceclofenac Cmax,ss | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Maximum concentration of drug in plasma at steady state
ilaprazole, aceclofenac AUCtau,ss | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Area under the plasma drug concentration-time curve within a dosing interval (tau) at steady state

SECONDARY OUTCOMES:
ilaprazole, aceclofenac Tmax,ss | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Time to maximum plasma concentration at steady state
ilaprazole, aceclofenac CLss/F | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Apparent clearance of drug in plasma at steady state
ilaprazole, aceclofenac Vdss/F | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Apparent volume of distribution at steady state
ilaprazole, aceclofenac Cmin,ss | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  Minimum concentration of drug in plasma at steady state
ilaprazole, aceclofenac fluctuation | Predose(0hour), after dose 0.5hour, 0.75hour, 1hour, 1.5hours, 2hours, 2.5hours, 3hours, 3.5hours, 4hours, 5hours, 6hours, 8hours, 10hours, 12hours
  fluctuation

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No